CLINICAL TRIAL: NCT01279278
Title: Does the Invitation by the General Practitioner Improve Patients' Participation in Colorectal Cancer Screening? A Cluster Randomised Controlled Study.
Brief Title: Does the Invitation by the General Practitioner Improve Patients' Participation in Colorectal Cancer Screening?
Acronym: Pagedocc1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: Adeca 75 (Other); Société de Formation Thérapeutique du Généraliste (Other); Hotel Dieu Hospital (Other)
Responsible Party: Pr Serge Gilberg, Université Paris Descartes - Département de Médecine Générale
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PAGEDOCC1
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2010-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Screening; General Practitioner; Fecal Occult Blood Tests
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
  Interventions: Other: Classical Letter
- Co-signed Letter (Experimental)
  Interventions: Other: Co-signed letter

INTERVENTIONS:
Other: Co-signed letter — Patients receive a personalized letter co-signed by their general practitioner and the medical coordinator of ADECA.
  Arms: Co-signed Letter
Other: Classical Letter — Patients receive classical letter signed by the coordinator doctor of ADECA
  Arms: Control

SUMMARY:
The propose of this study is to assess the effect of general practitioner's involvement on first patients' solicitation in screening for colorectal cancer by testing for faecal occult blood (FOBT).

ELIGIBILITY:
Inclusion Criteria:

* Aged : 50 to 74 years.
* Not having ever been invited to participate in colorectal screening.

Exclusion Criteria:

* Patients who have a Fecal Occult Blood Test for less than 2 years or a colonoscopy within the past 5 years or excluded for medical reasons (according to information known from ADECA).

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Completion of Fecal Occult Blod Test | 7 months
  Increased number of patients who completed the test for faecal occult blood following the first solicitation with the letter co-signed by general practitioner, compared with the conventional solicition(including replies exclusions).

SECONDARY OUTCOMES:
Measure the impact of co-signing on deadline for completion of the test after the mailing. | 7 months
Compare the proportion of uninterpretable tests. | 7 months
Compare the rate of completion of colonoscopy after a positive test (information received by ADECA in the follow-up), according to the specifications. | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Université Paris Descartes, Paris, Île-de-France Region, France